CLINICAL TRIAL: NCT00538109
Title: An Open-Label, Multicenter, Expanded Access Study of Oral AMN 107 in Adult Patients With Imatinib (Glivec®/Gleevec®_ - Resistant or Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC #2071-008
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: CML in Blast Crisis; Accelerated Phase oe Chronic Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

INTERVENTIONS:
Drug: Glivec®/Gleevec® — Chemotherapy

SUMMARY:
An Open-Label, Multicenter, Expanded Access Study of Oral AMN 107 in Adult Patients with Imatinib (Glivec®/Gleevec®_ - Resistant or Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase

ELIGIBILITY:
Inclusion Criteria:

* Patients with Imatinib (Glivec/Gleevec) Resistant or Intolerant CML in Blast Crisis, Accelerated Phase or Chronic Phase

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness | overall

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Chaudhri, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center